CLINICAL TRIAL: NCT02738086
Title: Physical Activity Behavior Change for Older Veterans After Dysvascular Amputation
Brief Title: Physical Activity Behavior Change for Older Adults After Dysvascular Amputation
Acronym: PABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: F2054-P
Record Dates: First submitted 2016-03-16; First posted 2016-04-14 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Amputation; Diabetes Mellitus, Type 2; Peripheral Artery Disease
Keywords: Amputation; Physical Activity; Rehabilitation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Peripheral Arterial Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early PABC Intervention (Experimental): GROUP 1 will participate in the Physical Activity Behavior Change (PABC) intervention phase during the first 3 months. GROUP 1 will then participate in a non-exercise control phase during the second 3 months.
  Interventions: Behavioral: Physical Activity Behavior Change (PABC)
- Wait-List Control Intervention (Experimental): GROUP 2 will participate in a non-exercise control phase during the first 3 months. GROUP 2 will then participate in the Physical Activity Behavior Change (PABC) intervention phase in the second 3 months.
  Interventions: Behavioral: Physical Activity Behavior Change (PABC)

INTERVENTIONS:
Behavioral: Physical Activity Behavior Change (PABC) — Home-based weekly sessions (30 min) using behavior change methods for promoting physical activity. Sessions will occur using home-based computer tablets for real-time video interface between the participant and therapist. Participants will wear wrist-mounted activity sensors with direct physical activity feedback during the intervention period to allow for behavioral feedback and action planning.
Behavioral: Physical Activity Behavior Change (PABC) — Home-based weekly sessions (30 min) using behavior change methods for promoting physical activity. Sessions will occur using home-based computer tablets for real-time video interface between the participant and therapist. Participants will wear wrist-mounted activity sensors with direct physical activity feedback during the intervention period to allow for behavioral feedback and action planning

SUMMARY:
This pilot study will use mobile-health technology to deliver an intervention designed for lasting physical activity behavior change. The study will assess the feasibility of using the Physical Activity Behavior Change(PABC) intervention for Veterans with lower limb amputation. This intervention will be delivered using wrist-worn wearable activity sensors and a home-based tablet computer to allow real-time physical activity feedback and video interface between the participants and the therapist.

DETAILED DESCRIPTION:
This pilot study will assess the feasibility of using the Physical Activity Behavior Change(PABC) intervention for Veterans with dysvascular lower limb amputation. In addition, preliminary efficacy of the PABC intervention will be assessed using a two-group randomized cross-over design. Testing will occur at baseline (pre-intervention), three months (end of intervention), and six months. The primary aim is to determine feasibility of using the PABC intervention with Veterans who have dysvascular amputation by measuring:

1. participant retention
2. dose goal attainment
3. participant acceptability
4. safety The secondary aim is to preliminary assess efficacy of the PABC intervention by measuring accelerometer-based physical activity and self-report disability effect sizes.

ELIGIBILITY:
Inclusion Criteria:

* Lower limb amputation 1-5 years prior to enrollment
* Type 2 Diabetes Mellitus and/or
* Peripheral Artery Disease
* Ambulatory using a lower limb prosthesis
* English speaking

Exclusion Criteria:

* Traumatic or cancer-related etiology of the lower limb amputation
* Unstable heart condition, including:

  * unstable angina
  * uncontrolled cardiac dysrhythmia
  * acute myocarditis
  * acute pericarditis
* Uncontrolled hypertension
* Acute systemic infection
* Prisoner
* Decisionally challenged volunteers
* Cancer
* Recent cerebral vascular accident (within two years)
* lower extremity wound or ulcer that limits ability to ambulate

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cory L. Christiansen, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christiansen CL, Miller MJ, Kline PW, Fields TT, Sullivan WJ, Blatchford PJ, Stevens-Lapsley JE. Biobehavioral Intervention Targeting Physical Activity Behavior Change for Older Veterans after Nontraumatic Amputation: A Randomized Controlled Trial. PM R. 2020 Oct;12(10):957-966. doi: 10.1002/pmrj.12374. Epub 2020 May 6. PMID 32248638

RESULTS

PARTICIPANT FLOW:
Groups:
- Early PABC Intervention (Months 1-3): GROUP 1 will participate in the Physical Activity Behavior Change (PABC) intervention phase during the first 3 months. GROUP 1 will then participate in a non-exercise control phase during the second 3 months.
  Physical Activity Behavior Change (PABC): Home-based weekly sessions (30 min) using behavior change methods for promoting physical activity. Sessions will occur using home-based computer tablets for real-time video interface between the participant and therapist. Participants will wear wrist-mounted activity sensors with direct physical activity feedback during the intervention period to allow for behavioral feedback and action planning.
- Wait-List Control Intervention (Months 4-6): GROUP 2 will participate in a non-exercise control phase during the first 3 months. GROUP 2 will then participate in the Physical Activity Behavior Change (PABC) intervention phase in the second 3 months.
  Physical Activity Behavior Change (PABC): Home-based weekly sessions (30 min) using behavior change methods for promoting physical activity. Sessions will occur using home-based computer tablets for real-time video interface between the participant and therapist. Participants will wear wrist-mounted activity sensors with direct physical activity feedback during the intervention period to allow for behavioral feedback and action planning.
Period: Overall Study
Arm/Group | Early PABC Intervention (Months 1-3) | Wait-List Control Intervention (Months 4-6)
Started | 16 | 15
Completed | 14 | 13
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early PABC Intervention | Wait-List Control Intervention | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (6.2) | 63.4 (8.9) | 65.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 15 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 12 | 14 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 15 | 31
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27 (5) | 31 (6) | 29 (6)
Time Since Amputation (months) [Mean (Standard Deviation); unit: months] | 37 (41) | 36 (16) | 36 (31)
Level of Amputation [Count of Participants; unit: Participants]
  Transtibial | 14 | 12 | 26
  Transfemoral | 2 | 3 | 5
Geriatric Depression Scale score [Mean (Standard Deviation); unit: units on a scale] — Scores are on a scale of 0 to 15, with scores of 0 to 5 being normal. A score greater than 5 suggests depression.
  units on a scale | 4.1 (4.0) | 3.7 (3.8) | 3.9 (3.9)
Mini-Mental Status Examination score [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 30 with scores above 24 indicating normal cognition.
  units on a scale | 28.4 (4.5) | 29.0 (1.6) | 28.7 (3.1)
Chakrabarty Grade score [Mean (Standard Deviation); unit: units on a scale] — Scoring system of residual-limb quality. Scores can range from -115 to 100. Higher scores indicate better residual limb quality.
  units on a scale | 84.8 (18.4) | 85.7 (12.4) | 85.2 (15.4)
Functional Comorbidity Index score [Mean (Standard Deviation); unit: Number of Comorbidities] — Scores can be between 0 and 18. Higher scores indicate a larger number of comorbidities.
  Number of Comorbidities | 6.8 (3.3) | 6.0 (3.2) | 6.4 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Retention Rate
Description: Retention rate will be measured as the percent of participants enrolled in the intervention who complete the intervention.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- GROUP 2: Wait-List Control Intervention: GROUP 2 will participate in a non-exercise control phase during the first 3 months. GROUP 2 will then participate in the Physical Activity Behavior Change (PABC) intervention phase in the second 3 months.
  Physical Activity Behavior Change (PABC): Home-based weekly sessions (30 min) using behavior change methods for promoting physical activity. Sessions will occur using home-based computer tablets for real-time video interface between the participant and therapist. Participants will wear wrist-mounted activity sensors with direct physical activity feedback during the intervention period to allow for behavioral feedback and action planning.
Arm/Group | Early PABC Intervention | GROUP 2: Wait-List Control Intervention
Number analyzed (Participants) | 16 | 15
Participants | 14 | 13

2. Primary Outcome: Dose Goal Attainment
Description: Dose goal attainment will be measured as the percent of participants in the intervention phase of the study who meet the dose goal of an average 3% increase in daily steps.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- PABC Intervention: Groups 1 and 2
  Physical Activity Behavior Change (PABC): Home-based weekly sessions (30 min) using behavior change methods for promoting physical activity. Sessions will occur using home-based computer tablets for real-time video interface between the participant and therapist. Participants will wear wrist-mounted activity sensors with direct physical activity feedback during the intervention period to allow for behavioral feedback and action planning.
Arm/Group | PABC Intervention
Number analyzed (Participants) | 29
Participants | 3

3. Primary Outcome: Acceptability
Description: Acceptability will be measured using the mean score of the Intrinsic Motivation Inventory - Interest / Enjoyment Subscale. The scores range from 1 to 7, with higher numbers indicating higher acceptability, and a null value of 5.0.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PABC Intervention
Number analyzed (Participants) | 29
score on a scale | 5.8 (0.8)

4. Primary Outcome: Study-Related Adverse Events
Description: Safety will be assessed as differences in rates of study-related adverse events between GROUP 1 and GROUP 2 during the first three months, when GROUP 1 is in the intervention phase and GROUP 2 is in the non-intervention control phase.
Time Frame: 3 months
Measure: Number; unit: Adverse Events
Arm/Group | Early PABC Intervention | GROUP 2: Wait-List Control Intervention
Number analyzed (Participants) | 16 | 15
Adverse Events | 20 | 29

5. Secondary Outcome: Accelerometer-Based Physical Activity
Description: Physical activity counts will be measured using a waist-mounted accelerometer-based physical activity monitor (Actigraph). The outcome will be average daily physical activity counts.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Steps
Arm/Group | Early PABC Intervention | GROUP 2: Wait-List Control Intervention
Number analyzed (Participants) | 14 | 13
Steps | 1609 [826 to 2393] | 1897 [1242 to 2551]

6. Secondary Outcome: Late Life Function and Disability Scale, Frequency
Description: The Late Life Function and Disability Scale (LLFDSI) will be used to assess the participant-reported disability at each test point. Scores range from 0 to 100, with higher scores indicating higher disability.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Early PABC Intervention | GROUP 2: Wait-List Control Intervention
Number analyzed (Participants) | 15 | 15
score on a scale | 49.3 [46.2 to 52.4] | 54.5 [48.5 to 60.6]

7. Secondary Outcome: Accelerometer-Based Physical Activity
Description: as for outcome 5
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Steps
Arm/Group | Early PABC Intervention | GROUP 2: Wait-List Control Intervention
Number analyzed (Participants) | 14 | 13
Steps | 1716 [948 to 2483] | 1773 [1189 to 2357]

8. Secondary Outcome: Late Life Function and Disability Scale, Frequency
Description: as for outcome 6
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Early PABC Intervention | GROUP 2: Wait-List Control Intervention
Number analyzed (Participants) | 14 | 13
score on a scale | 52.5 [48.6 to 56.3] | 51.3 [48.4 to 54.3]

9. Secondary Outcome: Late Life Function and Disability Scale, Limitation
Description: as for outcome 6
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Early PABC Intervention | GROUP 2: Wait-List Control Intervention
Number analyzed (Participants) | 15 | 15
score on a scale | 71.4 [63.2 to 79.7] | 68.1 [55.3 to 80.9]

10. Secondary Outcome: Late Life Function and Disability Scale, Limitation
Description: as for outcome 6
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Early PABC Intervention | GROUP 2: Wait-List Control Intervention
Number analyzed (Participants) | 14 | 13
score on a scale | 74.3 [65.3 to 83.3] | 68.6 [60.7 to 76.4]

ADVERSE EVENTS:
Time Frame: For Group 1 adverse event data were collected weekly during the 12 week intervention, and at 24 weeks. For Group 2 adverse event data were collected weekly during the 12 week attention control period and weekly during the 12 week intervention.
Groups:
- GROUP 1: Early PABC Intervention (Months 1-3): GROUP 1 will participate in the Physical Activity Behavior Change (PABC) intervention phase during the first 3 months. GROUP 1 will then participate in a non-exercise control phase during the second 3 months.
  Physical Activity Behavior Change (PABC): Home-based weekly sessions (30 min) using behavior change methods for promoting physical activity. Sessions will occur using home-based computer tablets for real-time video interface between the participant and therapist. Participants will wear wrist-mounted activity sensors with direct physical activity feedback during the intervention period to allow for behavioral feedback and action planning.
- GROUP 1: No Contact Phase (Months 4-6): GROUP 1 will participate in the Physical Activity Behavior Change (PABC) intervention phase during the first 3 months. GROUP 1 will then participate in a non-exercise control phase during the second 3 months.
- GROUP 2: PABC Attention Control (Months 1-3): GROUP 2 will participate in a non-exercise control phase during the first 3 months. GROUP 2 will then participate in the Physical Activity Behavior Change (PABC) intervention phase in the second 3 months.
- GROUP 2: PABC Intervention (Months 4-6): GROUP 2 will participate in a non-exercise control phase during the first 3 months. GROUP 2 will then participate in the Physical Activity Behavior Change (PABC) intervention phase in the second 3 months.
  Physical Activity Behavior Change (PABC): Home-based weekly sessions (30 min) using behavior change methods for promoting physical activity. Sessions will occur using home-based computer tablets for real-time video interface between the participant and therapist. Participants will wear wrist-mounted activity sensors with direct physical activity feedback during the intervention period to allow for behavioral feedback and action planning.
Arm/Group | GROUP 1: Early PABC Intervention (Months 1-3) | GROUP 1: No Contact Phase (Months 4-6) | GROUP 2: PABC Attention Control (Months 1-3) | GROUP 2: PABC Intervention (Months 4-6)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/16 | 2/16 | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 8/16 | 5/16 | 8/15 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GROUP 1: Early PABC Intervention (Months 1-3) (N=16) | GROUP 1: No Contact Phase (Months 4-6) (N=16) | GROUP 2: PABC Attention Control (Months 1-3) (N=15) | GROUP 2: PABC Intervention (Months 4-6) (N=15)
Cardiac Disorder - Other (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-Healing Wounds (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GROUP 1: Early PABC Intervention (Months 1-3) (N=16) | GROUP 1: No Contact Phase (Months 4-6) (N=16) | GROUP 2: PABC Attention Control (Months 1-3) (N=15) | GROUP 2: PABC Intervention (Months 4-6) (N=15)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 5 (5) | 3 (3)
Wound (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT02738086/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT02738086/ICF_001.pdf